**Study Title:** The Effects of Respiratory Training on Voice

**NCT #:** NCT04710862

**Document Title:** Statistical Analysis Summary

**Document Date:** May 25, 2025

Distribution characteristics were determined for all outcome measures to derive descriptive statistics and to test for statistical modeling assumptions (SPSS version 27.0 software). Pre- to post-training group differences and within-participant differences at follow-up timepoints were determined using mixed linear models to account for the effects of group, assessment timepoint, and timepoint x group interactions as well as correlated (repeated) measurements. Post-hoc tests for within-group comparisons of the long-term follow-up timepoints in the Respiratory Lung Volume Training (RLVT) condition were performed using a Sidak correction. Non-parametric tests or data transformation techniques were implemented for any variables that did not show normal distributions. Pre-training (baseline) equivalence of mean values between the RLVT and control training (CT) groups was tested through t-tests for all outcome measures. An alpha level of .05 defined statistical significance, and two-tailed tests were used for all tests.